CLINICAL TRIAL: NCT01658917
Title: Prospective Procurement of Solid Tumor Tissue to Identify Novel Therapeutic Targets
Brief Title: Collecting Solid Tumor Tissue to Identify New Treatments
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120175; 12-C-0175
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Cancer; Liver Cancer; Pancreatic Cancer; Melanoma
Keywords: Tissue Acquisition; Natural History
MeSH Terms: conditions — Gastrointestinal Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary: Patients greater than or equal to 18 years of age who have premalignant, primary or metastatic solid tumors based upon either radiographic or biochemical testing, or histological/cytological analysis

SUMMARY:
Background:

The NCI Surgery Branch has developed experimental therapies that involve taking white blood cells from patients' tumor or from their blood, growing them in the laboratory in large numbers, and then giving the cells back to the patient.

Objective:

This study will allow tissue samples obtained during the protocol screening process to be used for future and ongoing research in the NCI Surgery Branch

Eligibility:

Patients must meet the minimum eligibility criteria for an NCI surgery Branch Treatment Protocol

Design

Patients will undergo testing and evaluations as required by the appropriate NCI Surgery Branch Treatment protocol

DETAILED DESCRIPTION:
BACKGROUND:

* Recent advances and insights into the molecular pathogenesis of cancer have led to the development of novel molecular and biologic targeted therapies for the treatment of advanced cancer patients. A critical challenge in extending these studies involves the identification and validation of new therapeutic targets for future cancer therapies.
* The Surgery Branch, NCI has an interest in identifying novel molecular and biologic targets to facilitate the development of future cancer therapies. In addition, we have the primary responsibility for providing surgical consultative services to the NIH. As such, we are uniquely positioned to acquire and perform important studies on solid tumor tissue to help identify therapeutic targets that may have significant clinical ramifications.

OBJECTIVES:

- Primary Objective: To collect biologic samples from patients undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors for the purpose of identifying novel molecular and biologic therapeutic targets

ELIGIBILITY:

* Patients >= 18 years of age with radiographic evidence of, biochemical evidence of, or histologically/cytologically proven solid neoplasms who require diagnostic or therapeutic intervention as a part of the diagnosis and /or standard of care treatment and/or follow up for their neoplasm
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to planned intervention

DESIGN:

* A tissue acquisition trial in which tissues will be obtained at the time of intervention
* Tissue and blood will be processed at the time of collection, stored and then transferred to Dr. Rosenberg s laboratory for further processing.
* No investigational therapy will be given.
* It is anticipated that 1000 patients will be enrolled over a period of ten years

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must be greater than or equal to 18 years of age.
* Patients who have a premalignant, primary or metastatic solid tumors based upon either radiographic or biochemical testing, or histological/cytological analysis that requires surgery or biopsy as a part of the standard of care diagnosis, treatment and/or follow up.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.
* Patients must be planning to undergo surgery or biopsy as part of their treatment plan. Note: Patients will not be enrolled exclusively for the procurement of tissue samples.
* Patients who agree to undergo leukapheresis must meet the following criteria:
* Seronegative for HIV
* Seronegative for hepatitis B surface antigen and seronegative for

antibody to hepatitis C.

- CBC within normal limits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects greater than or equal to 18 years of age from both gender groups and all racial/ethnic groups who are undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors@@@
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
To collect biologic samples from patients undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors. | At time of surgery or biospy
  To collect biologic samples from patients undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors for the purpose of identifying novel molecular and biologic therapeutic targets.

SECONDARY OUTCOMES:
To collect detailed history, demographic, treatment data, and perioperative findings. | At time of consent
  To collect detailed history, demographic, treatment data, and perioperative findings in order to categorize and track the specific procedures and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Longo DL. Tumor heterogeneity and personalized medicine. N Engl J Med. 2012 Mar 8;366(10):956-7. doi: 10.1056/NEJMe1200656. No abstract available. PMID 22397658
- [Background] Yachida S, Jones S, Bozic I, Antal T, Leary R, Fu B, Kamiyama M, Hruban RH, Eshleman JR, Nowak MA, Velculescu VE, Kinzler KW, Vogelstein B, Iacobuzio-Donahue CA. Distant metastasis occurs late during the genetic evolution of pancreatic cancer. Nature. 2010 Oct 28;467(7319):1114-7. doi: 10.1038/nature09515. PMID 20981102
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0175.html